CLINICAL TRIAL: NCT04595227
Title: Glaucoma Screening Using Dynamic Analysis of Computerized Pupillary Light Reflex Assessment Device Via Iris Recognition Techniques
Brief Title: Glaucoma Screening Using Dynamic Analysis of Computerized Pupillary Light Reflex Assessment Device
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Chun Zhang, professor, Peking University
Other Study IDs: IRB00006761-M2020269
Record Dates: First submitted 2020-10-10; First posted 2020-10-20 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Primary Open Angle Glaucoma; Primary Open-Angle Glaucoma, Unspecified Eye; Primary Open Angle Glaucoma of Both Eyes; Suspect Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Normal Subjects: Healthy eyes had intraocular pressure of less than 22 mmHg with no history of increased intraocular pressure and normal standard automated perimetry (SAP) results.
  Interventions: Device: Computerized pupillary light reflex assessment device
- Suspect Glaucoma: Eyes with suspect glaucoma were defined as those with suspicious neuroretinal rim thinning or retinal nerve fiber layer (RNFL) defects on masked stereophotographic assessment, without repeatable abnormal SAP results. Eyes with suspect glaucoma also included those with intraocular pressure (IOP) > 21 mm Hg but with healthy-appearing optic discs and without repeatable abnormal SAP results
  Interventions: Device: Computerized pupillary light reflex assessment device
- Primary Open Angle Glaucoma, early stage: Eyes were classified as glaucomatous if they had repeatable (≥2 consecutive) abnormal SAP(Humphrey) test results or progressive glaucomatous changes on masked grading of stereophotographs, with or without abnormal SAP results. Abnormal SAP results were defined by a pattern standard deviation outside the 95% confidence limits or glaucoma hemifield test results outside the reference range.( -0.01dB≤MD≤-6.00dB)
  Interventions: Device: Computerized pupillary light reflex assessment device
- Primary Open Angle Glaucoma, moderate stage: Eyes were classified as glaucomatous if they had repeatable (≥2 consecutive) abnormal SAP(Humphrey) test results or progressive glaucomatous changes on masked grading of stereophotographs, with or without abnormal SAP results. Abnormal SAP results were defined by a pattern standard deviation outside the 95% confidence limits or glaucoma hemifield test results outside the reference range.( -6.01≤MD≤-12.00dB)
  Interventions: Device: Computerized pupillary light reflex assessment device
- Primary Open Angle Glaucoma, advanced stage: Eyes were classified as glaucomatous if they had repeatable (≥2 consecutive) abnormal SAP(Humphrey) test results or progressive glaucomatous changes on masked grading of stereophotographs, with or without abnormal SAP results. Abnormal SAP results were defined by a pattern standard deviation outside the 95% confidence limits or glaucoma hemifield test results outside the reference range.( -12.00≤MD≤-20.00dB)
  Interventions: Device: Computerized pupillary light reflex assessment device

INTERVENTIONS:
Device: Computerized pupillary light reflex assessment device — CPLRAD may serve as an effective screening tool for glaucomatous optic neuropathy, since they can dynamically detect abnormal pupillary responses from a novel sequence of light stimuli and functionally-shaped stimuli. CPLRAD can collect the clinical examination data and objectively measure the pupil dynamic parameters monocularly and/or binocularly as indicators from the retina and optic nerve in glaucoma patients.

SUMMARY:
To explore an effective diagnostic tool of glaucoma through the dynamic analysis of computerized pupillary light reflex assessment device (CPLRAD) pupillography based on iris recognition techniques and investigate its feasibility in glaucoma screening.

DETAILED DESCRIPTION:
Glaucoma is the leading cause of irreversible blindness worldwide, which is characterized by progressive loss of retinal ganglion cells (RGCs) and their optic nerve axons. Early diagnosis and treatment can effectively prevent the progression of the disease and avoid blindness. The damage of RGCs appears in the early stage of glaucoma, and the asymmetry of the eyes has also been observed clinically. CPLRAD may serve as an effective screening tool for glaucomatous optic neuropathy, since they can dynamically detect abnormal pupillary responses from a novel sequence of light stimuli and functionally-shaped stimuli. The current theoretical evidence of relative afferent pupillary defect/pupillary light reflex (RAPD/PLR) as a functional test for predicting nerve damage is insufficient, and pupil detection technology is not yet mature. Therefore, the investigators want to complete these tasks: 1) collect the clinical examination data and objectively measure the pupil dynamic parameters monocularly and/or binocularly as indicators from the retina and optic nerve in glaucoma patients 2) design RAPD/PLR detection technology and develop dynamic analysis system; 3) verify the feasibility of RAPD/PLR applied to early glaucoma screening through clinical trials. The pupil image dynamic analysis and iris recognition system will provide a simple, inexpensive and non-invasive screen tool, and is highly reliable and cost-effective.

ELIGIBILITY:
Inclusion Criteria:

* with open angles on gonioscopy
* best-corrected visual acuity ≥0.5
* spherical refraction within ±6.0 diopters (D), and cylinder correction within 3.0 D

Exclusion Criteria:

* eyes with any evidence of physical abnormality of the iris or pupils on slit-lamp examination
* eyes with a history of trauma or inflammation
* undergone an intraocular surgery or laser within the previous 6 months /except uncomplicated cataract surgery
* using systemic or topical medications that could affect pupil responses, including pilocarpine or atropine
* presence of any media opacities that prevented good quality optical coherence tomography (OCT) or fundus images
* presence of any retinal or neurological disease other than glaucoma abnormal ocular motility that prevents binocular fixation (eg, nystagmus, strabismus)
* with severe system diseases or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants are recruited from patients visiting at the Ophthalmologic Center of Peking University Third Hospital and from the general population through advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Constriction Velocity in One Eye in Different Groups | The test of each participant will complete the all procedures within 1 hour.
  The maximum constriction velocity will be calculated by the software
Maximum Dilation Velocity in One Eye in Different Groups | The test of each participant will complete the all procedures within 1 hour.
  The maximum dilation velocity will be calculated by the software.
Pupil Constriction Amplitude(ratio) in One Eye in Different Groups | The test of each participant will complete the all procedures within 1 hour.
  The pupil constriction amplitude(ratio) will be calculated by the software.
Baseline Pupil Size in One Eye in Different Groups | The test of each participant will complete the all procedures within 1 hour.
  The baseline pupil size is measured before the stimulus on.
Baseline Pupil Size(BPZ) Asymmetry between Two Eyes in Different Groups | The test of each participant will complete the all procedures within 1 hour.
  Asymmetry is calculated by a formula:
  RAPD score of BPZ= 10 * log10 (baseline pupil size in right eye/baseline pupil size in left eye)
Maximum Constriction Velocity(MCV) Asymmetry between Two Eyes in Different Groups | The test of each participant will complete the all procedures within 1 hour.
  Asymmetry is calculated by a formula:
  RAPD score of MCV= 10 * log10 (maximum constriction velocity in right eye/maximum constriction velocity in left eye)
Maximum Dilation Velocity(MDV) Asymmetry between Two Eyes in Different Groups | The test of each participant will complete the all procedures within 1 hour.
  Asymmetry is calculated by a formula:
  RAPD score of MDV = 10 * log10 (maximum dilation velocity in right eye/maximum dilation velocity in left eye)
Pupil Constriction Amplitude(ratio) Asymmetry between Two Eyes in Different Groups | The test of each participant will complete the all procedures within 1 hour.
  Amplitude(ratio) is calculated by: (DIAMETER resting-DIAMETER constricted) / DIAMETER resting
  Asymmetry was calculated by a formula:
  RAPD score of Amplitude = 10 * log10 (pupil constriction amplitude in right eye/pupil constriction amplitude in left eye)

CONTACTS AND LOCATIONS:
Overall Officials: Chun Zhang, MD/PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hosipital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No